CLINICAL TRIAL: NCT06790810
Title: Observational Study on Dynamic Changes of Blood Pressure During Post-epileptic Seizure Stage: A Multicenter Study
Brief Title: Observational Study on Dynamic Changes of Blood Pressure During Post-epileptic Seizure Stage (OCBPS)
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Fujian Medical University Union Hospital (Other); The First Hospital of Hebei Medical University (Other); Henan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); General Hospital of Ningxia Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shandong Provincial Hospital (Other Government); Ruijin Hospital Luwan Branch (Other); Shenzhen University General Hospital (Other); Beijing Sanbo Brain Hospital (Other); Xuanwu Jinan Hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial) (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Other Study IDs: 2024-322-002
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy; Seizure; Blood Pressure
Keywords: Seizures; epilepsy; blood pressure; change; post-seizure; post-epileptic seizure stage
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This article details a multicenter study on changes of blood pressure and heart rate during post-epileptic seizure stage.

DETAILED DESCRIPTION:
In contrast to the well-documented changes in heart rate and respiration, post-seizure changes in blood pressure have received insufficient attention. Fluctuations in blood pressure may worsen brain injury and elevate the risk of Sudden Unexpected Death in Epilepsy (SUDEP), yet evidence regarding postictal blood pressure changes remains limited.

This multicenter study aims to investigate the changes of blood pressure and heart rate during post-epileptic seizure stage in epilepsy patients, providing high-quality evidence on postictal hemodynamic changes and laying the foundation for future interventions. The study will enroll 2000 seizure events from hospitalized epilepsy patients aged 14-80 years between October 2024 and October 2025. Data on blood pressure, heart rate and blood oxygen will be collected during multiple time intervals post-seizure, alongside clinical information such as seizure type, duration, and medication use.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-80 years old, male and female;
2. Meet the diagnostic criteria for epilepsy, including focal epilepsy and generalized epilepsy.
3. Patients diagnosed with epilepsy, with at least one seizure during the hospitalization.
4. Seizures lasting longer than 30 seconds (including convulsive and non-convulsive status epilepticus, if seizure cessation can be determined and medications were recorded, they can be included).
5. Hypertensive patients who are on antihypertensive medication and have well-controlled blood pressure are eligible.
6. Patients who agree to participate in the study.

Exclusion Criteria:

1. Patients with structural heart disease, coronary artery disease (CAD), cardiomyopathy
2. Patients with severe systemic diseases
3. Pregnancy
4. Preictal seizures or myoclonic seizures.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient epilepsy patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of baseline blood pressure versus post-epileptic seizure blood pressure (systolic and diastolic) | within 1 hour
  Baseline blood pressure and blood pressure measurements (systolic and diastolic) immediately after seizure (0-1 minute), at 3 minutes (2-4 minutes), 5 minutes (4-6 minutes), 10 minutes (9-11 minutes), 20 minutes (19-21 minutes), 30 minutes (29-31 minutes), and 60 minutes (59-61 minutes) post-seizure.

SECONDARY OUTCOMES:
Comparison of baseline heart rate versus post-epileptic seizure heart rate | within 1 hour
  Baseline heart rate and heart rate measurements immediately after seizure (0-1 minute), at 3 minutes (2-4 minutes), 5 minutes (4-6 minutes), 10 minutes (9-11 minutes), 20 minutes (19-21 minutes), 30 minutes (29-31 minutes), and 60 minutes (59-61 minutes) post-seizure.
Comparison of baseline blood-oxygen versus post-epileptic seizure blood-oxygen | within 1 hour
  Baseline oxygen saturation and oxygen saturation measurements immediately after seizure (0-1 minute), at 3 minutes (2-4 minutes), 5 minutes (4-6 minutes), 10 minutes (9-11 minutes), 20 minutes (19-21 minutes), 30 minutes (29-31 minutes), and 60 minutes (59-61 minutes) post-seizure.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Liankun Ren, MD, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No